CLINICAL TRIAL: NCT03763630
Title: Primary Prevention of Atopy and Asthma With House Dust Mite Sublingual Immunotherapy: 6-8 Years Follow up
Brief Title: MAPS & ITEC Cohorts: 6-8 Years Follow-up
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Isle of Wight NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Southampton CHI0808
Record Dates: First submitted 2018-11-22; First posted 2018-12-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Immunotherapy; Allergy and Immunology; Asthma
Keywords: Atopy; Early childhood; House Dust-mite; Sublingual immunotherapy
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Active Comparator): House dust-mite SLIT
  Interventions: Drug: House dust-mite SLIT
- Control arm (Placebo Comparator): Normal saline
  Interventions: Drug: Normal saline
- Observation cohort (No Intervention): ITEC observational cohort, no intervention administered

INTERVENTIONS:
Drug: House dust-mite SLIT — received 2000 standard treatment units of glycerinated HDM allergen extract (ALK-AbellÓ) per day. Normal saline was administered to the placebo group. 11 µg of HDM allergen (equal parts of Dermatophagoides pteronyssinus and Dermatophagoides farinae) administered twice daily as oral drops.
  Other Names: glycerinated HDM allergen extract (ALK-AbellÓ)
  Arms: Intervention arm
Drug: Normal saline — Normal saline administered in same frequency and manner as intervention
  Other Names: Normal saline placebo control
  Arms: Control arm

SUMMARY:
This study represents the follow-up, age 6-8 years, of children recruited at birth into two cohorts. The first cohort, the Mite Allergen Prevention Study (MAPS) was a double-blind, randomized controlled trial of the use of house dust-mite immunotherapy in the primary prevention of atopy and asthma. The Immune Tolerance in Early Childhood (ITEC) cohort is a separate observational cohort following up infants at high risk of atopy and correlating atopic disease development with epigenetic markers.

DETAILED DESCRIPTION:
There is an epidemic of allergic disease in childhood and current preventative strategies have failed to demonstrate effectiveness outside of isolated trials. In a previous study, the efficacy of sublingual immunotherapy (SLIT) with house dust mite in preventing the development of allergic sensitisation in infants was assessed. The long term objective was to assess the effect of the intervention on the subsequent development of asthma. The hypothesis is that high dose oral immunotherapy will induce immune tolerance and reduce development of allergic sensitisation and later clinical asthma and allergy. A total of 111 infants at high risk of allergy (with ≥2 first degree relatives affected by asthma or allergy) but with no evidence of allergic sensitisation at recruitment were recruited. These infants were randomised at 6 months of age to receive a year of active HDM (House dust-mite) allergen extract delivered as SLIT or placebo intervention. At 18 months of age, there was a significant reduction in cumulative allergic sensitisation in the SLIT intervention group and a trend for reduction in allergic symptoms. They have also been followed up at 3 years of age. The data currently being analysed.

Additionally, an observational cohort (Immune Tolerance in Early Childhood, ITEC) was recruited at birth with the same inclusion criteria as the interventional one and assessed in the same way up to 3 years. This cohort has provided additional control data and samples to utilise in the analyses.

This proposed study is the 6-8 year follow up of these interventional and observational cohorts. The aim of the 6-8 year assessment is to assess the efficacy of prophylactic oral immunotherapy with HDM allergen in preventing the later development of asthma. The hypothesis is that high dose oral immunotherapy will induce immune tolerance and reduce development of allergic sensitisation and later clinical asthma and allergy. Participants will be assessed 6-8 years after finishing the intervention. The assessment will include a questionnaire, skin prick testing to the common aeroallergens and food allergens and lung function. Families and study investigators will both be blinded to participants' original treatment allocations. An additional aim is to investigate the epigenetic and immune mechanisms involved in the development of asthma and allergy and how allergen immunotherapy influence this process.

ELIGIBILITY:
Inclusion Criteria:

•Inclusion in original study cohorts at birth

•≥2 first-degree relatives with allergic disease (food allergy, asthma, eczema, rhinoconjunctivitis)

Exclusion Criteria:

* Not included in the original study cohorts
* Skin-prick test positive to any allergen (HDM, cat, grass pollen, peanut, egg and milk) age 5 months

Ages: 5 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 263 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Clinical Asthma - parental questionnaire | Age 6 years
  Comparison of clinical asthma, as assessed by parental questionnaire, at age 6 years between control and intervention groups. Clinical asthma will be defined as either doctor diagnosed asthma or presence of wheeze and asthma medication use within the past year.
Clinical Asthma- spirometry with reversibility | 6 years
  Comparison of clinical asthma, as assessed by lung function testing, at age 6 years between control and intervention groups. Clinical asthma will be defined as in improvement in FEV1 (Forced Expiratory Volume in 1 second) of 12% or more following administration of salbutamol inhaler (bronchodilator).

SECONDARY OUTCOMES:
Bronchial hyper-responsiveness | Age 6 years
  Comparison of bronchial hyperresponsiveness, as determined by methacholine bronchial allergen challenge, at age 6 years.
Asthma comparison | Age 6 years
  Comparison of asthma, as defined by wheeze plus bronchial hyperreactivity
Airway inflammation level- exhaled nitric oxide measurement | Age 6 years
  Comparison of airway inflammation level, as assessed by exhaled nitric oxide, between placebo and intervention group age 6 years
Cumulative sensitization | Age 6 years
  Comparison of cumulative sensitization to one or more of 6 common allergens, as assessed by skin prick test, up to 6-8 years of age between control and interventions groups.
Cumulative aeroallergen sensitization | Age 6 years
  Comparison of cumulative sensitization to one or more of 6 common aeroallergens, as assessed by skin prick test, up to 6-8 years of age between control and interventions groups.
House dust-mite sensitization | Age 6 years
  Comparison of sensitization to house dust mite, as assessed by skin prick test, at 18 months, 3 years and 6-8 years of age between control and intervention groups.
Clinical atopic disease- parental questionnaire | Age 6 years
  Comparison of clinical allergic diseases/symptoms (atopic eczema, wheeze, allergic rhinitis, food allergy) at 18 months, 3 years and 6 years of age between control and intervention groups. Presence of clinical disease evaluated through parental questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Graham Roberts, Prof, Principal Investigator — University of Southampton
Locations (2):
- United Kingdom (2):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - David Hyde Asthma and Allergy Centre, Newport, Isle of White

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zolkipli Z, Roberts G, Cornelius V, Clayton B, Pearson S, Michaelis L, Djukanovic R, Kurukulaaratchy R, Arshad SH. Randomized controlled trial of primary prevention of atopy using house dust mite allergen oral immunotherapy in early childhood. J Allergy Clin Immunol. 2015 Dec;136(6):1541-1547.e11. doi: 10.1016/j.jaci.2015.04.045. Epub 2015 Jun 12. PMID 26073754